CLINICAL TRIAL: NCT05329285
Title: CABG or PCI in Patients With Ischemic Cardiomyopathy - A Randomized Registry Clinical Trial
Brief Title: CABG or PCI in Patients With Ischemic Cardiomyopathy
Acronym: STICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Region Örebro County (Other); Karolinska University Hospital (Other); University Hospital, Umeå (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPM dnr 2021-04972
Record Dates: First submitted 2022-03-17; First posted 2022-04-15 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
Keywords: PCI; CABG
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: An open-label, multicentre randomized registry trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Coronary Intervention (PCI) (Experimental): Patients will be revascularized by PCI
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI)
- Coronary artery bypass grafting (CABG) (No Intervention): Patients will be revascularized by CABG

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI) — Alternative treatment
  Arms: Percutaneous Coronary Intervention (PCI)

SUMMARY:
The STICH-SWEDEHEART trial will compare PCI vs CABG for revascularization of patients with HF and LV systolic dysfunction (LV ejection fraction (LVEF) <40%) and multi-vessel coronary artery disease.

DETAILED DESCRIPTION:
Short background/ Rationale/Aim:

CABG has been shown to prolong survival in patients with reduced left ventricular (LV) function and multi-vessel coronary artery disease and "CABG is recommended as the ﬁrst revascularization strategy choice in patients with multi-vessel disease and acceptable surgical risk". However, a major concern with CABG is the early risk of complications, including death and stroke. Although PCI has lower rates of peri-procedural complications than CABG in patients without heart failure (HF), this has not been confirmed in patients with HF. The lack of contemporary data comparing CABG and PCI in HF leaves clinicians with no guidance as to which option to choose, and a robust trial is therefore necessary. The STICH-SWEDEHEART trial will compare PCI vs CABG for revascularization of patients with HF and LV systolic dysfunction (LV ejection fraction (LVEF) < 40%) and multi-vessel coronary artery disease.

Study objective:

To test whether PCI is non-inferior to CABG for revascularization of patients with ischemic heart failure.

Study design:

Multicentre, open-label, randomized controlled trial

Study population:

Patients with ischemic cardiomyopathy and reduced ejection fraction.

Number of subjects:

470 subjects

Investigational treatment:

PCI

Treatment in control group:

CABG

Study endpoints:

Primary endpoint (variable):

The occurrence of the composite of death, stroke, non-procedural myocardial infarction or heart failure hospitalization at 3 years.

Key secondary endpoint The hierarchical occurrence (in descending order of importance) at 3-year follow-up of time to death, time to stroke, time to non-procedural myocardial infarction, number of heart failure hospitalizations and 1-year Kansas City Cardiomyopathy Questionnaire (KCCQ) score; evaluated using the win ratio approach.

Secondary safety endpoints

In-hospital occurrence of the following:

1. Death
2. Stroke
3. Non-procedural myocardial infarction
4. The occurrence of in-hospital BARC ≥3 bleeding

   Time to the occurrence of the following:
5. Mediastinitis
6. Pericardial tamponade Other secondary endpoints

1. Time to the occurrence of the following: A. Death, stroke or non-procedural myocardial infarction B. Death or heart failure hospitalization C. Heart failure hospitalization D. Coronary revascularization E. Death or myocardial infarction F. Death or stroke 2. Total number of days in-hospital during index hospitalization 3. Total number of days in intensive care unit during index hospitalization 4. Quality of life at 30 days and 365 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Symptomatic HF defined as NYHA HF class II-IV within 1 month of enrolment
3. LVEF ≤ 40% quantified by either echocardiography or gated SPECT ventriculography, or magnetic resonance (MR) or any other recognized assessment of LVEF
4. Meaningful amount of myocardium at risk because of CAD (BCIS myocardial jeopardy score ≥ 6 on a recent (> 6 months) coronary angiogram);
5. Heart team believes that a meaningful revascularization can be achieved by both PCI or CABG, with complete revascularization defined as residual ischemia in <10% of the left ventricle
6. Heart team agrees that guideline directed medical therapy (GDMT) has been initiated for ≥1 month in prevalent and newly diagnosed cases. In patients hospitalized with newly diagnosed iLVSD (with or without acute coronary syndrome (ACS)) requiring revascularization before discharge, GDMT needs to be initiated, when possible, in-hospital before randomization, with the expectation that it will be titrated to maximally tolerated doses after revascularization
7. Written informed consent obtained

Exclusion Criteria:

1. Previous randomization in the study
2. Decompensated heart failure requiring inotropic /adrenergic support, invasive or non-invasive ventilation or intra-aortic balloon pump/ventricular assist device therapy less than 48 hours prior to randomization
3. Recent (<1 month) type 1 myocardial infarction
4. Recent PCI (<3 months)
5. Valvular heart disease or any other cardiac conditions (e.g. LV aneurysm) requiring surgical repair/replacement
6. Prohibitive bleeding risk or clinical scenario mandating avoidance of long-term dual antiplatelet therapy
7. Expected survival less than 3 years due to non-cardiac illness
8. Circumstances likely to lead to poor treatment compliance
9. Individuals for whom record in public health databases is not accessible (non-eligibility to public health system, parallel healthcare systems
10. Pregnancy or woman of childbearing potential who is not sterilized or using a medically accepted form of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2052-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac event | 3 years
  The occurrence of the composite of death, stroke, non-procedural myocardial infarction or heart failure hospitalization

SECONDARY OUTCOMES:
The occurrence of death | 3 years
  Time to death
The occurrence of stroke | 3 year
  Time to stroke
The occurrence of non-procedural myocardial infarction, | 3 year
  Time to non-procedural myocardial infarction,
The occurrence of heart failure hospitalizations | 3 year
  Number of heart failure hospitalizations
Kansas City Cardiomyopathy Questionnaire (KCCQ) score | 1 year
  Kansas City Cardiomyopathy Questionnaire score; evaluated using the win ratio approach. High score mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Kardiologen, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thuan PQ, Chuong PTV, Nam NH, Dinh NH. Coronary Artery Bypass Surgery: Evidence-Based Practice. Cardiol Rev. 2025 Jul-Aug 01;33(4):344-351. doi: 10.1097/CRD.0000000000000621. Epub 2023 Dec 19. PMID 38112423